CLINICAL TRIAL: NCT06340919
Title: Hearing Aid Algorithms for Sudden Sounds
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Oticon (Unknown)
Responsible Party: Principal Investigator, AlexanderLab, Associate Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1406014978-241
Record Dates: First submitted 2024-03-24; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Control (No Intervention): Each participant will listen to recordings of sentences processed by a hearing aid with settings for treating sudden sounds set to OFF.
- Low Sudden Sound Reduction (Experimental): Each participant will listen to recordings of sentences processed by a hearing aid with settings for treating sudden sounds set to Low.
  Interventions: Device: Sudden Sound Reduction Setting
- High Sudden Sound Reduction (Experimental): Each participant will listen to recordings of sentences processed by a hearing aid with settings for treating sudden sounds set to High.
  Interventions: Device: Sudden Sound Reduction Setting
- Maxiumum Sudden Sound Reduction (Experimental): Each participant will listen to recordings of sentences processed by a hearing aid with settings for treating sudden sounds set to Maximum.
  Interventions: Device: Sudden Sound Reduction Setting

INTERVENTIONS:
Device: Sudden Sound Reduction Setting — Each participant will listen to recordings of sentences processed by a hearing aid with settings for treating sudden sounds set to Low, High, or Maximum. Recordings with the different settings will be randomized from trial to trial.
  Arms: High Sudden Sound Reduction; Low Sudden Sound Reduction; Maxiumum Sudden Sound Reduction

SUMMARY:
This study explores the impact of hearing aid settings for managing sudden sounds on speech comprehension and recall in individuals with hearing loss. Participants will undergo a comprehensive audiological evaluation, case history, and cognitive assessments. Subsequently, they will participate in listening experiments designed to measure sentence recognition, storage, and retrieval under various sudden sound reduction conditions recorded through a hearing aid. The experiment will be complemented by subjective preference ratings to identify participant comfort and listening clarity associated with different sudden sound reduction settings.

DETAILED DESCRIPTION:
Participants will first undergo a comprehensive audiologic test battery and questionnaires. The audiologic test battery will consist of (a) pure tone audiometry: basic and extended high frequency, (b) tympanometry, (c) wideband acoustic immittance, (d) acoustic reflexes, and (e) otoacoustic emissions. They will also complete online questionnaires at home: (a) loudness and annoyance, (b) noise exposure, (c) general survey concerning hearing in difficult situations, medical and otologic history, noise exposure, tinnitus, balance, sensory sensitivity (lights, sound, touch, smell, taste), and amplification. In addition, they will complete online tests of temporal gap detection.

Participants who meet the study inclusion criteria (hearing aid candidacy based on air conduction thresholds between 2000 and 6000 Hz) will return to the lab for two additional sessions. During the first session, before starting the main experiment, they will complete the Working Memory Questionnaire (Vallat-Azouvi et al., 2012), which evaluates short-term storage, attention, and executive control. The first main experiment evaluates sentence recognition, storage, and retrieval. Participants will hear two sentences in a row: one by a male or female talker and the other by a person of the opposite gender. Participants are asked to remember the first sentence while listening to the second sentence. They will be asked to repeat the last sentence aloud (a measure of sentence recognition). Then, they will be asked to type the first sentence (a measure of sentence storage and retrieval). Most, but not all, sentences will have sudden soft sounds and one sudden loud sound. Participants will hear each pair of sentences only once; they will not be allowed to replay the audio.

Sentence pairs were recorded through hearing aids in an anthropomorphic manikin with one of four treatments for sudden sounds: (1) off, (2) low, (3) high, and (4) maximum. Participants will listen to 36 sentence pairs for each of the four treatments. All will contain sudden soft sounds (e.g., keyboard typing, footsteps, chewing, etc.) throughout the two sentences; half will contain a sudden loud sound (e.g., gunshot, door slamming, iPhone notification, etc.) at the onset of a keyword in the first sentence and the other half in the second sentence. Control stimuli do not contain sudden sounds. Conditions assigned to each sentence list (18 pairs) will be randomly assigned to each sentence participant. In addition, all stimuli were recorded using one of eight standardized audiometric configurations. Participants will listen to the recordings made with the audiogram that best matches the hearing loss in one of their ears. Participants can scale the overall output up or down 15 dB to accommodate differences in loudness preferences. Finally, all recordings were filtered before playback to remove the resonance associated with the external ear properties of the anthropomorphic manikin using the test earphones.

Participants will return to the lab for a second session in which they will rate their preferences for the different sudden sound reduction settings. Before beginning the experiment, they will complete the Visual Letter Monitoring (VLM) test (Gatehouse et al., 2003). The VLM test assesses attention, reaction time, continuous performance, and working memory capabilities. Participants will observe letters displayed one at a time in large font on a computer screen. Letters will switch between vowels and consonants in an unbroken sequence with intervals of 2 ("slow") or 1 second ("fast"). Participants will press the space bar on the computer keyboard or a button on the touchscreen whenever three sequential letters (Consonant-Vowel-Consonant) form a word.

For the subjective preference portion of the experiment, participants listen to sentences recorded with two different sudden sound reduction settings (6 combinations comprised of off, low, high, or maximum). Each sentence will be played twice, in succession, but with different pairs of settings from trial to trial. Following each trial, they will select which setting they prefer overall. Additionally, they will choose the setting they favor more for the speech (identified as the clearest, most natural, and least distorted) and the setting they favor for the noise (deemed the most comfortable, least annoying, and softest). To indicate their preference, participants will press the "1" button if the first setting was more to their liking or the "2" button if they found the second setting superior. Participants are permitted to revise their choice and switch their selection. They can re-listen to the sentence pairing as many times as needed. Participants will listen to 72 sentences for each combination of settings to provide sufficient power to conduct single-subject statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Air conduction thresholds 25-70 dB HL from 2000 - 6000 Hz
* Native English speakers

Exclusion Criteria:

* Retrocochlear hearing loss

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech recognition | Through study completion, on average 2 hours
  Number of keywords repeated from a sentence just heard
Recall | Through study completion, on average 2 hours
  Number of keywords repeated from a sentence heard previously
Preference | Through study completion, on average 2 hours
  Paired comparison, preference ratings

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Alexander, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data stored as a CSV file will be shared. Individual participants' responses to each trial (audio recording) will be provided.
Time Frame: Upon formal acceptance of the published manuscript; to be stored indefinitely.
Access Criteria: Open
URL: https://purr.purdue.edu/